CLINICAL TRIAL: NCT01602081
Title: Ligation of the Intersphincteric Fistula Tract With Tissue Graft Placement for Treatment of Persistent Trans-sphincteric Anal Fistula
Brief Title: Ligation of the Intersphincteric Fistula Tract (LIFT) + Biodesign for Anal Fistula
Acronym: LIFT+Graft
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-012
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Anal Fistula
Keywords: Anal fistula; Ligation of the intersphincteric fistula tract; LIFT; Tissue graft
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- LIFT+Biodesign
  Interventions: Device: reinforce soft tissue

INTERVENTIONS:
Device: reinforce soft tissue — reinforce soft tissue

SUMMARY:
The LIFT+Biodesign® study is a post-market observational study to evaluate the rate of fistula closure in patients with persistent trans-sphincteric anal fistula who receive the Biodesign® Tissue graft as part of their LIFT procedure.

ELIGIBILITY:
Inclusion Criteria:

* Persistent primary or recurrent trans-sphincteric anal fistula

Exclusion Criteria:

* Patients with prior fistulotomy, fistulectomy, LIFT, cutting seton or advancement flap procedure
* Fistula with multiple tracts
* Recto-vaginal fistula
* Active infection in the anal fistula
* Physical allergies or cultural objections to porcine products
* Patient is not medically fit to undergo the LIFT procedure as judged by the treating physician
* Previous diagnosis of collagen disorder
* History of Crohn's Disease, Irritable Bowel Syndrome, radiation therapy in the rectoanal region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regional and Community Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Closure of the anal fistula | 6 months

SECONDARY OUTCOMES:
Closure of the anal fistula | 12 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California Irvine, Orange, California
  - Rush University Medical Center, Chicago, Illinois
  - Indiana University Hospitals, Indianapolis, Indiana
  - Kendrick Regional Center, Indianapolis, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Mount Sinai Hospital, New York, New York
  - Case Medical Center, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania